CLINICAL TRIAL: NCT02395328
Title: The Impact of Future's Families Orphans and Vulnerable Children Home Visiting Program in Tshwane Townships of South Africa
Brief Title: Home Visiting for OVC in Tshwane Townships of South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Social Work (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tonya Renee Thurman, Principle Investigator, Associate Professor, Tulane University School of Social Work
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AID-674-A-12-00002-FFGS
Record Dates: First submitted 2015-03-05; First posted 2015-03-23 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: HIV
Keywords: Orphans and vulnerable children (OVC); Home visiting intervention; South Africa; Program evaluation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care worker home visitation (Experimental): Care Workers provide biweekly home visits and offer residing caregivers and children information and psychosocial support, and encourage their awareness and accessing of external health and social services.
  Interventions: Behavioral: Care Worker Home Visitation
- Wait List (No Intervention): Access to homework classes are made available to all participants' children at schools supported by the implementing organization.

INTERVENTIONS:
Behavioral: Care Worker Home Visitation — Primary services include biweekly home visits from Care Workers trained, mobilized and supported by Futures Families, a South African non-government organization working to support OVC in six townships within the greater Tshwane area (also known as Pretoria) of South Africa.
  Arms: Care worker home visitation

SUMMARY:
This study consists of a one-year randomized controlled trial investigating the impact of mobilized care workers trained and supported by Futures Families, a South African non-profit organization, that provide biweekly home visits to families with orphans and vulnerable children (OVC) in Tshwane (aka Pretoria) townships, South Africa. Future Families takes a family-based approach to addressing the needs of OVC by providing caregivers with information, psychosocial support, and access to external services. Caregivers will participate in a survey providing information on their personal wellbeing as well as key indicators reflecting the wellbeing of each child under their care. Newly enrolled caregivers will be randomly assigned to either program participation beginning in late 2014 or to delayed participation following the impact survey about one year later. The data will be used to test for changes in a set of key program indicators pertaining to child protection, HIV prevention, psychosocial wellbeing, education and early childhood development. This study aims to strengthen the evidence base for effective family centered programming to address the needs of HIV-affected children and their caregivers.

DETAILED DESCRIPTION:
With an estimated 5.6 million people living with HIV in South Africa, the AIDS epidemic has led to a large number of orphaned or otherwise vulnerable children (OVC) and families. Both psychosocial challenges and economic hardship are disproportionately common in homes where an orphan or HIV-infected adult resides. OVC caregivers may suffer emotional distress, have limited social support and experience family discord. Research reports a heightened risk of mental health problems among OVC caregivers, including grandparents and HIV positive parents. Addressing the needs of OVC caregivers is integral to a comprehensive, family-based approach. OVC programming principles therefore emphasize the importance of interventions that endeavor to enhance the psychosocial well-being and caregiving capacity of OVC guardians.

The purpose of this study is to evaluate the impact of Future Families Care Worker home visiting program. Future Families is a South African non-government organization working in six townships located within the greater Tshwane area (also known as Pretoria) of South Africa. Future Families trains and mobilizes Care Workers from the local community to provide biweekly home visits to OVC households to offer caregivers and children information, psychosocial support, and encourage awareness and accessing of health and social services.

Future Families will identify an approximate 500 eligible beneficiaries families between May-July 2014. These families are randomly assigned to receive a Care Worker beginning in August 2014 or approximately 12 months later following the second survey. Random assignment will be accomplished using computer software designed for random allocation of subjects to groups, and interviewers will be blind to individuals' group assignments. Both groups of newly-enrolled beneficiaries will be offered homework assistance classes at a Future Families facility, to ensure that even the control group receives some benefit from enrolment.

In each of these homes, data will be collected from the adult caregiver, the adult in the home who has primary responsibility for the care of residing children in June-July 2014 and again in November 2015 (following an approximate one year of service delivery). Further, we also obtained data from 282 current adult caregiver beneficiaries from within the same communities who have been enrolled in the program for at least one year, to facilitate an immediate post-test assessment, comparing the wellbeing of these current beneficiaries with newly enrolled beneficiaries. The post-test is designed to provide insight into potential impact of past efforts as well as potential areas for improvement. This information is particularly useful at the outset of the evaluation as it can inform and direct program implementation to address gaps while bolstering areas of success.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over at the time of study enrollment;
* Enrolled in a selected Future Families site;
* Willing and able to consent to study participation

Exclusion Criteria:

* Are not able to give informed consent due to known or recognizable cognitive or psychiatric impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in access to HIV testing services indicator | Baseline, 12 months post-intervention
  Percent of children and guardians (reported separately) who have ever been tested for HIV and received most recent test results
Change in psychosocial wellbeing indicator | Baseline, 12 months post-intervention
  Multi-item indicator to determine the percent of guardians with basic social support and the percent of guardians with high levels of negative feelings;
Change in early childhood development indicators | Baseline, 12 months post-intervention
  Multi-item indicator to determine the percent of children 1-5 years who are fully immunized; Percent of children <5 years of age who recently engaged in stimulating activities with any household member over 15 years of age and percent of children age 1-5 enrolled in a crèche or other early childhood development centre.
Change in school attendance indicator | Baseline, 12 months post-intervention
  Percent of school-age children attending school regularly.
Change in access to social services indicators | Baseline, 12 months post-intervention
  Percent of children with a verified birth certificate or other identity documentation and percent of eligible children and caregivers receiving grants.

SECONDARY OUTCOMES:
Change in household economics indicator | Baseline, 12 months post-intervention
  Multi-item indicator to determine the percent of children whose basic material needs are met; percent of children with needed school supplies; percent of households earning income (other than from grants) for the past 3 months; percent of guardians currently earning income (other than from grants); percent of households with moderate or severe hunger; and percent of households with a member in a savings group;
Change in health status indicator | Baseline, 12 months post-intervention
  Multi-item indicator to determine the percent of children and guardians (reported separately) too sick to participate in daily activities in past 14 days; percent of guardians with high levels of daily functioning; percent of households with a male who has been circumcised; and the percent of HIV positive children and guardians adhering to an ARV regimen.
Change in harsh punishment practices indicator | Baseline, 12 months post-intervention
  Percent of guardians who used corporal punishment on any child in the household in the past 3 months

OTHER OUTCOMES:
Demographics and Background indicator | Baseline, 12 months post-intervention
  Multi-item indicator to determine the percent of children who have been orphaned (single/double/maternal/paternal can be reported separately); percent of children living without a biological parent in the home; percent of children living with a chronic illness; percent of children living with someone who is chronically ill; percent of children living in child or youth-headed households; percent of children whose primary guardian is age 60 or older; average child-adult ratio for households; percent of guardians who are likely AIDS-sick (three or more symptoms); and percent of guardians subject to stressful experiences in the last year.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya R Thurman, PhD MPH, Principal Investigator — Tulane University School of Social Work

IPD SHARING:
Plan to Share IPD: Undecided